CLINICAL TRIAL: NCT06730412
Title: ctDNA Liquid Biopsy for Early Assessment of Residual Disease in HPV-associated Head and Neck Cancer (Clear-HPVca)
Acronym: Clear-HPVca
Status: Completed | Type: Observational
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH); National Institutes of Health (NIH) (NIH); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Daniel L. Faden, MD, Assistant Professor, Harvard Medical School, Massachusetts General Hospital
Other Study IDs: 18-653; R03DE030550 (NIH)
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2024-12

CONDITIONS: HPV Positive Oropharyngeal Squamous Cell Carcinoma
Keywords: MRD; HPV; HPV+ HNSCC; NGS; HPV-DeepSeek; squamous cell carcinoma; head and neck squamous cell carcinoma; circulating tumor DNA; liquid biopsy; minimal residual disease
MeSH Terms: conditions — Carcinoma, Squamous Cell; Squamous Cell Carcinoma of Head and Neck; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, plasma, and tumor tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HPV-associated head and neck cancer patients treated with surgery: AJCC 8 Stage I-III HPV+ head and neck cancer patients treated with curative intent surgery

SUMMARY:
The purpose of this study is to test a new liquid biopsy assay for detecting residual disease after surgery in patients with HPV-associated head and neck cancer.

DETAILED DESCRIPTION:
Human papillomavirus associated head and neck squamous cell carcinoma (HPV+HNC) is the most common HPV-associated cancer in the United States. Surgery is a common approach for primary treatment of early-stage HPV+HNC. Many patients who undergo surgery receive adjuvant radiation or chemoradiation therapy to treat potential residual disease, which is currently predicted based on clinicopathologic risk factors including positive margins, extranodal extension, multiple positive lymph nodes, vascular invasion, and lymphatic invasion. However, there are limitations in predicting residual disease based on the use of these features alone - the use of clinicopathologic risk factors for prediction is non-standardized and has poor individualized predictive and prognostic capacity. Currently, there are no established biomarkers to predict residual disease.

Circulating tumor DNA (ctDNA) is an emerging minimally invasive prognostic biomarker, for detecting molecular residual disease (MRD) and predicting recurrence in multiple solid cancers. Prospective trials in cancers such as colorectal cancer have demonstrated not only strong Disease Free Survival (DFS) prognostic capacity but also Overall Survival (OS). Previous studies have demonstrated that HPV+HNCs release circulating tumor HPV DNA (ctHPVDNA) into the blood where it serves as an accurate real-time biomarker of disease status after surgery. In patients without pathological risk factors, ctHPVDNA is rapidly cleared after surgery. In patients with residual disease, ctHPVDNA remains elevated after surgery. However, initial studies have showed that patients with microscopic levels of residual disease are often not detected by current approaches using droplet digital PCR (ddPCR), suggesting significantly more sensitive assays are necessary.

HPV-DeepSeek is an HPV whole genome next-generation sequencing assay which is significantly more sensitive than ddPCR-based approaches. The investigators aim to conduct a prospective observational cohort study of HPV+HNC patients treated with curative intent surgery to test the primary hypothesis that patients with MRD detection after surgery will have inferior 2-year DFS and OS and the secondary hypothesis that patients with MRD detection after treatment completion (surveillance) will have inferior 2-year DFS and OS.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Newly diagnosed, untreated, histologically confirmed HPV-associated head and neck cancer
* Scheduled for curative intent resection as primary treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-2

Exclusion Criteria:

* Not meeting all inclusion criteria
* Pregnant
* Receiving treatment for concurrent second malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AJCC 8 Stage I-III HPV+ Head and Neck Cancer patient undergoing curative intent surgical resection
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-10-31 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 2 years
  Disease free survival in patients with versus without minimal residual disease detection after surgery
Overall survival | 2 years
  Overall survival in patients with versus without minimal residual disease detection after surgery

SECONDARY OUTCOMES:
Disease free survival | 2 years
  Disease free survival in patients with versus without minimal residual disease detection after treatment completion
Overall survival | 2 years
  Overall survival in patients with versus without minimal residual disease detection after treatment completion

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Otolaryngology - Head and Neck Surgery, Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No